CLINICAL TRIAL: NCT01144403
Title: A Phase II Multicenter Open-label Study of MabThera(Rituximab) Addition to Regularly Prescribed Chemotherapy in Patients With Untreated Mantle Cell Lymphoma
Brief Title: A Study of MabThera (Rituximab) Addition to Regularly Prescribed Chemotherapy in Patients With Untreated Mantle Cell Lymphoma.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML22489; 2009-011433-27
Record Dates: First submitted 2010-06-14; First posted 2010-06-15 (Estimated); Results first posted 2016-08-29 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-07

CONDITIONS: Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Cyclophosphamide; fludarabine; Mitoxantrone; Rituximab

ARMS (1):
- Rituximab (Experimental): Rituximab, 375 milligram per meter square (mg/m^2) was given intravenously on Day 1 and then every 28 days (+/-7 days) for 6 cycles, followed by 2 consolidated infusions in responders as rituximab induction therapy. Rituximab infusions were administered concomitantly with prescribed chemotherapy i.e., fludarabine, cyclophosphamide and mitoxantrone (maximum 6 cycles).
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Mitoxantrone; Drug: Rituximab

INTERVENTIONS:
Drug: Cyclophosphamide — as prescribed, 6 cycles
Drug: Fludarabine — as prescribed, 6 cycles
Drug: Mitoxantrone — as prescribed, 6 cycles
Drug: Rituximab — 375 mg/m^2 intravenously, Day 1 of each 28-day cycle, up to 8 cycles
  Other Names: Mabthera/Rituxan

SUMMARY:
This multicenter, open-label study will assess the efficacy and safety of MabThera (rituximab) added to standard chemotherapy in participants with untreated Mantle Cell Lymphoma not eligible for autologous stem cell transplantation. Participants will receive MabThera (372 mg/m^2 intravenously) on Day 1 of each 28-day treatment cycle in addition to standard chemotherapy for 6 cycles. In participants experiencing complete or partial response, MabThera will be continued as consolidation therapy for 2 more cycles.

ELIGIBILITY:
Inclusion Criteria:

* adult participants, >/=18 years of age
* untreated Mantle Cell Lymphoma, not eligible for Autologous Stem Cell Transplantation
* known mantle cell lymphoma international prognostic index (MIPI) at diagnosis
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* adequate hematological, renal and hepatic function

Exclusion Criteria:

* known hypersensitivity to murine proteins or chemotherapy regimen
* previous first-line therapy
* history of other malignancy within the last 5 years, except for squamous cell carcinoma, basal cell carcinoma of the skin or in situ cervical carcinoma
* active infection
* clinically significant cardiac disease
* regular corticosteroid treatment in the 4 weeks prior to first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- Romania (6):
  - Brasov
  - Bucharest
  - Cluj-Napoca
  - Iași
  - Târgu Mureş
  - Timișoara

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total 8 participants were enrolled from Romania.
Groups:
- Rituximab: Rituximab, 375 milligram per meter square (mg/m^2) was given intravenously on Day 1 and then every 28 days (+/-7 days) for 6 cycles, followed by 2 consolidated infusions in responders as rituximab induction therapy. Rituximab infusions were administered concomitantly with prescribed chemotherapy i.e., fludarabine, cyclophosphamide and mitoxantrone (maximum 6 cycles).
  Cyclophosphamide: as prescribed, 6 cycles
  Fludarabine: as prescribed, 6 cycles
  Mitoxantrone: as prescribed, 6 cycles
  Rituximab [Mabthera/Rituxan]: 375 mg/m^2 intravenously, Day 1 of each 28-day cycle, up to 8 cycles
Period: Overall Study
Arm/Group | Rituximab
Started | 8
Completed | 3
Not Completed | 5
Not completed — Lost to Follow-up | 3
Not completed — Death | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Rituximab: Rituximab, 375 milligram per meter square (mg/m^2) was given intravenously on Day 1 and then every 28 days (+/-7 days) for 6 cycles, followed by 2 consolidated infusions in responders as rituximab induction therapy. Rituximab infusions were administered concomitantly with regularly prescribed chemotherapy i.e., fludarabine, cyclophosphamide and mitoxantrone (maximum 6 cycles).
  Cyclophosphamide: as prescribed, 6 cycles
  Fludarabine: as prescribed, 6 cycles
  Mitoxantrone: as prescribed, 6 cycles
  Rituximab [Mabthera/Rituxan]: 375 mg/m^2 intravenously, Day 1 of each 28-day cycle, up to 8 cycles
Arm/Group | Rituximab
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.50 (7.964)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Overall Response Rate (ORR) was determined by tumor response according to International Workshop Group to Standardize Response Criteria for mantle cell lymphoma (MCL) criteria from confirmed evaluations of both target, radiographically evaluated, and non-target lesions. A responder is defined as a subject experiencing either a complete (CR)/ unconfirmed complete (Cru), or partial response (PR) by these criteria. As per criteria; CR = disappearance of all evidence of disease; CRu = the sum of the product of the diameters (SPD) of multiple nodes decreased by at least 75%; PR = regression of measurable disease and no new sites.
Time Frame: Up to 50 months (approximately)
Population: Efficacy population included all the participants who had received at least one dose of study treatment.
Measure: Number; unit: percentage of participants
Groups:
- Rituximab: Rituximab, 375 milligram per meter square (mg/m^2) was given intravenously on day 1 and then every 28 days (+/-7 days) for 6 cycles, followed by 2 consolidated infusions in responders as rituximab induction therapy for mantle cell lymphoma. Rituximab infusions were administered concomitantly with regularly prescribed chemotherapy i.e., fludarabine, cyclophosphamide and mitoxantrone (maximum 6 cycles).
  cyclophosphamide: as prescribed, 6 cycles
  fludarabine: as prescribed, 6 cycles
  mitoxantrone: as prescribed, 6 cycles
  rituximab [Mabthera/Rituxan]: 375 mg/m^2 intravenously, day 1 of each 28-day cycle, up to 8 cycles
Arm/Group | Rituximab
Number analyzed (Participants) | 8
percentage of participants | 87.5

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as time from date of enrollment to the date of death, regardless of the cause of death.
Time Frame: From the time of enrollment until death due to any cause (up to 50 months [approximately])
Population: Efficacy population included all the participants who had received at least one dose of study treatment.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Rituximab
Number analyzed (Participants) | 8
days | 927 [0.000 to 2204.066]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the interval between the day of enrollment and the first documentation of progressive disease or death. Progression of disease is defined as at least a 20 percent (%) increase in the sum of longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of 1 or more new lesions.
Time Frame: From the time of enrollment until death due to any cause (up to 50 months [approximately])
Population: Efficacy population included all the participants who had received at least one dose of study treatment.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Rituximab
Number analyzed (Participants) | 8
days | 653 [537.058 to 768.942]

4. Secondary Outcome: Number of Participant With Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with study treatment.
Time Frame: Up to 50 months (approximately)
Population: Safety population included all the participants who had received at least one dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Rituximab
Number analyzed (Participants) | 8
participants | 8

ADVERSE EVENTS:
Time Frame: Up to approximately 50 months
Arm/Group | Rituximab
Serious Adverse Events (participants affected / at risk) | 3/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=8)
Pneumonia (Infections and infestations) | 1
Neutropenia (Infections and infestations) | 1
Toxicity (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=8)
Anemia (Blood and lymphatic system disorders) | 3
Leucopenia (Blood and lymphatic system disorders) | 4
Gastric Pain (Gastrointestinal disorders) | 1
Ascending Aorta Dilatation (Vascular disorders) | 1
Drug Eruption (Injury, poisoning and procedural complications) | 2
Dermatitis Eczematous (Skin and subcutaneous tissue disorders) | 1
Tracheitis (Respiratory, thoracic and mediastinal disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hepatitis Ag HBS+ (Hepatobiliary disorders) | 1
Herpes (Infections and infestations) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Vertiginous syndrome (Nervous system disorders) | 1
Supraventricular arrhythmia (Cardiac disorders) | 1
Respiratory Virosis (Respiratory, thoracic and mediastinal disorders) | 1
Oral Candidiasis (Infections and infestations) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 5
ß2-microglobuline ↗ (Blood and lymphatic system disorders) | 1
C- reactive protein (Blood and lymphatic system disorders) | 1

LIMITATIONS AND CAVEATS:
The study was prematurely terminated with 8 participants enrolled, all of them are included into the statistical analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.